CLINICAL TRIAL: NCT04033757
Title: A Population-based Cohort of Osteoarthritis: the Xiangya Osteoarthritis Study
Status: Active, not recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: University of Nottingham (Other); Harvard University (Other)
Responsible Party: Sponsor
Other Study IDs: 201510506
Record Dates: First submitted 2019-07-04; First posted 2019-07-26 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; cohort study; population-based
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Biospecimen Retention: Samples With DNA — Blood, urine, stool, saliva, dental plaque
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sub-cohort 1: 1,469 participants were enrolled in 2015. Three follow-ups have been completed in 2016, 2017, and 2020. They will be asked to participate in follow-up in 2023 and 2026.
- Sub-cohort 2: 1,267 participants were enrolled in 2018. They will be asked to participate in follow-up in 2021, 2024, 2027, and 2030.
- Sub-cohort 3: 1,340 participants were enrolled in 2019. They will be asked to participate in follow-up in 2022, 2025, 2028, and 2031.

SUMMARY:
The purpose of this study is to examine the natural history, phenotypes and risk factors of osteoarthritis (OA) and pain at different joints, and to examine the association between OA structure changes, inflammation and pain for knee and hand OA.

DETAILED DESCRIPTION:
Objectives:

1. To understand the natural history of osteoarthritis (OA) at different joints (knee, hip, hand, foot and lumbar).
2. To identify different phenotypes of OA (e.g., generalized OA, rapidly progressive knee and hand OA, tibiofemoral OA and patellofemoral OA), their association with pain (e.g., peripheral pain, central pain, nociceptive pain and neuropathic pain) and consequences.
3. To examine risk factors of OA (lifestyle habits, nutritional, metabolic, anatomical and genetic factors, etc.) at each joint as well as multiple joints.
4. To determine the association between x-ray structure change, ultrasound synovial changes and pain and other symptoms of OA at knee and hand joints within the large-sample community-based population.
5. To predict the progression of knee and hand OA within new-onset early-stage knee and hand OA patients, and to identify the rapidly progressive knee and hand OA phenotypes and their related risk factors.
6. To investigate the association between gut microbiota and OA.
7. To investigate the association between oral microbiota and OA.

Design: This is a prospective community-based cohort study.

Participants: Subjects included in this study were a randomly selected sample of residents, aged 50 years or older from rural mountainous communities of Longshan County, Hunan Province, China. 4000 people were planned to be recruited, divided into three sub-cohorts. 1,469 participants were enrolled in sub-cohort 1 in 2015, and two follow-ups have been completed in 2016 and 2017. 1,267 participants were enrolled in sub-cohort 2 in 2018. 1,340 participants were enrolled in sub-cohort 3 in 2019. Each sub-cohort will be followed every three years regularly.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years old or above
2. Residents of the randomly selected communities

Exclusion Criteria:

1. Inability to give informed consent
2. Terminal or mental illness
3. Pregnant women

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects included in this study were a randomly selected sample of residents, aged 50 years or older, from rural mountainous communities of Longshan County, Hunan Province, China.
Sampling Method: Probability Sample
Enrollment: 4080 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of multiple joints osteoarthritis. | At enrollment.
  Measured by radiographs of multiple joints.
Incidence of multiple joints osteoarthritis. | At 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by radiographs of multiple joints, and the incidence of osteoarthritis can be calculated at each follow-up time point.
Progression of multiple joints osteoarthritis. | At 3, 6, 9, 12 years follow-ups after enrollment.
  The changes of joint space and osteophytes are measured by radiographs of multiple joints, to assess the progression of multiple joints osteoarthritis.

SECONDARY OUTCOMES:
Ultrasound detected changes of knee, thigh muscle, and hand. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Ultrasound examination of both knee joints, quadriceps, hamstrings muscle and 15 peripheral joints of wrist and hand.
Changes of pain intensity of knee, hip, hand and lumbar. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by visual analog scale (VAS).
Changes of pain experience of knee. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by intermittent and constant osteoarthritis pain (ICOAP) questionnaire.
Changes of neuropathic pain of knee. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by painDETECT questionnaire (PDQ).
Changes of patient's belief about knee pain. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by illness perception questionnaire (IPQ).
Changes of pain catastrophizing of knee. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by pain catastrophizing scale (PCS).
Prevalence of knee/hip/patellofemoral joint pain. | At enrollment.
  Measured by a question that "In the past 12 months, have you had knee/hip/patellofemoral joint pain lasting most days of at least a month?"
Incidence of knee/hip/patellofemoral joint pain. | At 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by a question that "In the past 12 months, have you had knee/hip/patellofemoral joint pain lasting most days of at least a month?", and the incidence of knee/hip/patellofemoral joint pain can be calculated at each follow-up time point.
Changes of global assessment of knee and hip. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by the Western Ontario and McMaster Universities (WOMAC) score.
Changes of global hand function. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by the Functional Index for Hand Osteoarthritis (FIHOA).
Changes of pain-related disability of lumbar osteoarthritis. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by the Roland-Morris Disability Questionnaire (RMDQ).
Changes of the results of 30s repetition chair stand test. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  To test the ability to rise from a chair. Record the times a participant stand up and sit down from a chair within 30 seconds.
Changes of the results of 20-meter walk test. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Record the time a participant spent on walking for 20 meters.
Changes of the results of timed up and go test. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Record the time a participant to rise from a standard armchair, walk as quickly but as safely as possible distance of 3 meters, turn, walk back to the chair and sit down.
Changes of the results of standing balance test. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Record the score of standing balance using a standard test protocol. Tests of standing balance included full tandem, semi-tandem, and side-by-side stands.
Changes of grip strength. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by a Jamar Hydraulic Hand Dynamometer.
Changes of pinch strength. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by a Jamar Hydraulic Pinch Gauge.
Changes of quadriceps strength. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by a 'Nicholas Manual Muscle Tester' (Lafayette Instruments).
Changes of hamstrings strength. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by a 'Nicholas Manual Muscle Tester' (Lafayette Instruments).
Changes of hip abductor. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by a 'Nicholas Manual Muscle Tester' (Lafayette Instruments).
Changes of the results of squatting ability test. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  The squatting ability was evaluated by using a 1-4 scale (1 = full squat, no use of arms; 2 = full squat, arms used for support; 3= full squat, examiner assistance needed; 4 = attempted, unable to attain full squat).
Changes of the results of stair climbing test. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Record the time a participant to ascended and descended a flight of five 14 cm steps stair as quickly as possible.
Changes of the results of quantitative sensory testing. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by a hand-held pressure algometer (Wagner, FDIX25) .
Changes of the results of body composition analysis. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by a InBody 770 Body Composition Analyser.
Prevalence of nodal osteoarthritis. | At enrollment.
  Nodal osteoarthritis was determined using a validated line diagram and classified as present in those reporting nodes on at least two rays of both hands.
Prevalence of widespread pain. | At enrollment.
  A modified body pain mannequin with two questions on symptom severity and widespread pain index (2011 ACR criteria on fibromyalgia) was included to allow scoring of fibromyalgia as a diagnosis with binary (present/absent) classification using a validated tool.
Incidence of widespread pain. | At 3, 6, 9, 12 years follow-ups after enrollment.
  A modified body pain mannequin with two questions on symptom severity and widespread pain index (2011 ACR criteria on fibromyalgia) was included to allow scoring of fibromyalgia as a diagnosis with binary (present/absent) classification using a validated tool. The incidence of knee/hip/patellofemoral joint pain can be calculated at each follow-up time point.
Changes of physical and mental health. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by the 12-Item Short-Form Health Survey (SF-12).
Changes of sleep quality. | At enrollment, and 3, 6, 9, 12 years follow-ups after enrollment.
  Measured by the Medical Outcomes Study (MOS) Sleep Scale.
Prevalence of sarcopenia. | Every round of surveys since year 2018.
  Sarcopenia would be diagnosed according to the Asian Working Group for Sarcopenia 2019 algorithm.
Incidence of sarcopenia. | At 3, 6, 9, 12 years follow-ups after enrollment.
  Sarcopenia would be diagnosed according to the Asian Working Group for Sarcopenia 2019 algorithm. And the incidence of sarcopenia can be calculated at each follow-up time point.

CONTACTS AND LOCATIONS:
Overall Officials: Guanghua Lei, Doctor, Study Chair — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
This cohort study will collect different types of data. The amount of data is large. The investigators have not decided what specific data sets to be shared yet.

REFERENCES:
- [Derived] Zhu Y, Li J, Zhang Y, Zhang W, Doherty M, Yang Z, Cui Y, Zeng C, Lei G, Yang T, Wei J. Association between hyperuricaemia and hand osteoarthritis: data from the Xiangya Osteoarthritis Study. RMD Open. 2023 Dec 1;9(4):e003683. doi: 10.1136/rmdopen-2023-003683. PMID 38053456